CLINICAL TRIAL: NCT02330406
Title: Effect of Anagliptin and Sitagliptin on Low-density Lipoprotein Cholesterol in Patients With Type 2 Diabetes and Cardiovascular Risk Factors: Randomized Controlled Trial
Brief Title: Randomized Evaluation of Anagliptin Versus Sitagliptin On Low-density lipoproteiN Cholesterol in Diabetes Trial
Acronym: REASON
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institute for Clinical Effectiveness, Japan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ICE_2014_01R
Record Dates: First submitted 2014-12-30; First posted 2015-01-05 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Dipeptidyl-Peptidase 4 Inhibitors; LDL Cholesterol; Glycosylated Hemoglobin; Diabetes Mellitus; Coronary Disease
Keywords: Dipeptidyl-Peptidase 4 Inhibitors; LDL Cholesterol; Glycosylated Hemoglobin; Diabetes Mellitus; Coronary Disease
MeSH Terms: conditions — Diabetes Mellitus; Coronary Disease | interventions — anagliptin; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anagliptin (Active Comparator): Anagliptin 100 mg bid for 52 weeks. Can increase to 200 mg bid if needed.
  Interventions: Drug: Anagliptin
- Sitagliptin (Active Comparator): Sitagliptin 50 mg qd for 52 weeks. Can increase to 100 mg qd if needed
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: Anagliptin — Suiny 100 mg
  Other Names: Suiny
  Arms: Anagliptin
Drug: Sitagliptin — Januvia 50 mg Glactiv 50 mg
  Other Names: Januvia; Glactiv
  Arms: Sitagliptin

SUMMARY:
The purpose of this study is to determine whether Anagliptin or Sitagliptin are effective in reducing the low-density lipoprotein cholesterol in patients with type 2 diabetes and cardiovascular risk factors on statin.

DETAILED DESCRIPTION:
Diabetes is a significant cause of cardiovascular and cerebrovascular events. Especially, diabetic patients with cardiovascular risk factors were significantly higher risk for cardiovascular and cerebrovasculara event. Therefore, several medical management strategies including anti-diabetic medications and statins were considered for those patients. However, in spite of such treatment, still many patients have cardiovascular and cerebrovascular events. One of the hypothesis is the residual risk such as elevated low-density lipoprotein cholesterol (LDLC) even with statin therapy. Anagliptin, one of the dipeptidyl peptidase-4 (DPP4) inhibiors, was reported to reduce LDLC and may have pontential to decrease the cardiovascular and cerebrovascular risk for such patients on statins. We, thus, conduct a randomized controlled trial to compare Anagliptin or Sitagliptin in terms of change of LDLC for 52 weeks as well as glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes with cardiovascular risk factors (*) who treated with diet, exercise or antidiabetic medications
* Patients who were treated with statins for 8 weeks or longer
* Patients with low-density lipoprotein cholesterol equal to or greater than 100 mg/dL in the at least one of three measurements after the administration of statins
* Patients with glycerated hemoglobin (HbA1c, NGSP) equal to or greater than 6.0 % (7.0 % if patients were not treated with dipeptidyl-peptidase 4 inhibitors) and lesser than 10.5 %

(*) cardiovascular risk factors were any of following conditions

1. Presence of stenosis (>=25%) or plaque on the previous coronary angiography or coronary CT
2. Presence of coronary calcification on the previous coronary CT
3. History of acute coronary syndrome
4. History of percutaneous coronary intervention or coronary artery bypass graft
5. History of stroke (ischemic stroke or hemorrhagic stroke)
6. History of transient ischemic attack
7. History of peripheral artery diseases or aortic disorders
8. Ankle-Brachial Index (AMI) equal to or less than 0.9 in the past measurement
9. Presence of carotid artery plaque (including Max IMT >=1.1mm) on carotid ultrasonography in the past

Exclusion Criteria:

* Patients with type 1 diabetes
* Patients with triglyceride equal to or greater than 400 mg/dL in the previous fasting measurements
* Patients with pregnancy, possible pregnancy, or on breast-feeding
* Patients with severe infections, perioperative status, or severe trauma
* Patients with renal dysfunction (creatinine >= 2.4 mg/dl for men, >= 2.0 mg/dl for women)
* Patients who were received glucagon-like peptide-1receptor agonists
* Patients whom physician in charge considered inappropriate for the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 353 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Change in low-density lipoprotein cholesterol | 52-weeks
Change in glycated hemoglobin | 52-weeks

SECONDARY OUTCOMES:
Change in fasting glucose | 52-weeks
Change in fasting insulin | 52-weeks
Change in 1.5-Anhydro-D-glucitol | 52-weeks
Change in C peptide | 52-weeks
Change in total cholesterol, triglyceride, non high dencisty lipoprotein cholesterol | 52-weeks
Change in Apolipoprotein A1, Apolipoprotein B, Apolipoprotein E | 52-weeks
Change in Apolipoprotein B48 | 52-weeks
Change in small dense low density lipoprotein | 52-weeks
Change in high sensitivity C-reactive protein | 52-weeks
Change in interleukin-6 | 52-weeks
Change in cholesterol absorption marker (campesterol; sitosterol) | 52-weeks
Change in cholesterol synthesis marker (lathosterol) | 52-weeks
Change in high molecular weight adiponectin | 52-weeks
Change in ratio of albumin and creatinine in urine | 52-weeks
Progression, unchange, remission rate of microalbumin and macroalbumin in urine | 52-weeks
Change in estimated glomerular filtration rate | 52-weeks
Change in glycated hemoglobin stratified by body mass index and waist circumference | 52-weeks
Correlation between glycated hemoglobin and body mass index or waist circumference | 52-weeks
Change in intima-media thickness or flow mediated dilation | 52-weeks
Change in postprandial glucose, insulin and activated glucagon-like peptide-1 | 52-weeks
Change in lipid profile and molecular size measured | 52-weeks
Change in fatty acid fraction | 52-weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shinichiro Ueda, MD, PhD, Principal Investigator — Professor of Medicine, Department of Clinical Pharmacology & Therapeutics, University of the Ryukyus
Locations (1):
- Department of Cardiovascular Medicine, Tomishiro Central Hospital, Tomishiro, Okinawa, Japan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Furuhashi M, Sakuma I, Morimoto T, Higashiura Y, Sakai A, Matsumoto M, Sakuma M, Shimabukuro M, Nomiyama T, Arasaki O, Node K, Ueda S. Treatment with anagliptin, a DPP-4 inhibitor, decreases FABP4 concentration in patients with type 2 diabetes mellitus at a high risk for cardiovascular disease who are receiving statin therapy. Cardiovasc Diabetol. 2020 Jun 15;19(1):89. doi: 10.1186/s12933-020-01061-0. PMID 32539832
- [Derived] Chihara A, Tanaka A, Morimoto T, Sakuma M, Shimabukuro M, Nomiyama T, Arasaki O, Ueda S, Node K. Differences in lipid metabolism between anagliptin and sitagliptin in patients with type 2 diabetes on statin therapy: a secondary analysis of the REASON trial. Cardiovasc Diabetol. 2019 Nov 16;18(1):158. doi: 10.1186/s12933-019-0965-3. PMID 31733647
- [Derived] Morimoto T, Sakuma I, Sakuma M, Tokushige A, Natsuaki M, Asahi T, Shimabukuro M, Nomiyama T, Arasaki O, Node K, Ueda S. Randomized Evaluation of Anagliptin vs Sitagliptin On low-density lipoproteiN cholesterol in diabetes (REASON) Trial: A 52-week, open-label, randomized clinical trial. Sci Rep. 2019 Jun 12;9(1):8537. doi: 10.1038/s41598-019-44885-x. PMID 31189978
- [Derived] Ueda S, Shimabukuro M, Arasaki O, Node K, Nomiyama T, Morimoto T. Effect of Anagliptin and Sitagliptin on Low-Density Lipoprotein Cholesterol in Type 2 Diabetic Patients with Dyslipidemia and Cardiovascular Risk: Rationale and Study Design of the REASON Trial. Cardiovasc Drugs Ther. 2018 Feb;32(1):73-80. doi: 10.1007/s10557-018-6776-z. PMID 29435776